CLINICAL TRIAL: NCT03473275
Title: Central Blood Pressure Regulation by the Brainstem and Influence by Renal Sympathetic Afference: a Functional Magnetic Resonance Imaging (MRI) Study in Hypertensive and Normotensive Participants
Brief Title: Brain BOLD fMRI in Hypertensive and Normotensive Participants
Acronym: BRAIrdN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, PD Dr. Grégoire Wuerzner, Primary Investigator, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2018-00105
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension,Essential
Keywords: Sympathetic nervous system; Blood oxygen level dependent; Brainstem; Contrast enhanced ultrasound; Kidney function; Hypertension; Renal denervation
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma: cathecholamines, plasma renin activity (PRA), Aldosterone, Neuropeptide Y (NPY)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: control: Healthy normotensive participants. Cold pressor test on feet 3 times for 40 seconds during brain BOLD fMRI (2 runs), renal ultrasound and contrast-enhanced ultrasound.
  PinPrick test on feet 3 times for 40 seconds during brain BOLD fMRI (2 runs), renal ultrasound and contrast-enhanced ultrasound.
  Interventions: Diagnostic Test: Cold Pressor test; Diagnostic Test: PinPrick test
- 2: untreated hypertensive: Untreated (or off antihypertensive drugs) hypertensive patients (ABPM proven essential hypertension).
  Cold pressor test on feet 3 times for 40 seconds during BOLD fMRI (2 runs), renal ultrasound and contrast-enhanced ultrasound.
  Interventions: Diagnostic Test: Cold Pressor test
- 3. resistant hypertensive: Patients with proven resistant hypertension and not renal denervated or for whom a renal denervation is planned according to the criteria of the CHUV.
  Cold pressor test on feet 3 times for 40 seconds during BOLD fMRI (2 runs), renal ultrasound and contrast-enhanced ultrasound.
  Interventions: Diagnostic Test: Cold Pressor test
- 4. renal denervation: Patients with a renal denervation. Cold pressor test on feet 3 times for 40 seconds during BOLD fMRI (2 runs), renal ultrasound and contrast-enhanced ultrasound.
  Interventions: Diagnostic Test: Cold Pressor test

INTERVENTIONS:
Diagnostic Test: Cold Pressor test — Both feet in icy waterbath alternated with body temperature water
Diagnostic Test: PinPrick test — Pricking both feet with a needle using gravity (without penetrating) alternated with cotton swap
  Groups: 1: control

SUMMARY:
This study will explore the brainstem activity in response to stress in hypertensive patients and normotensive subjects. In addition, it will evaluate if the response in hypertensive patients can be modulated by blocking the afferent signalling of sympathetic nervous system from the kidney to the brain achieved by renal denervation.

The investigators hypothesize that the change in BOLD signal intensity in response to stress is higher in hypertensive patients than in normotensive subjects and that in patients responsive to renal denervation the change in BOLD signal intensity in response to stress is decreased compared to non-responders or to non-denervated resistant hypertensive patients.

DETAILED DESCRIPTION:
In hypertension, the overactivity of the sympathetic nervous system (SNS) has been found to be implicated in its initiation, maintenance and adverse consequences. The SNS is composed of an afferent and efferent arm, which brings sensory information to the brain (e.g. brainstem and hypothalamus) and transmits sympathetic outflow from the brain to the peripheral organs, respectively. Selective removal of the afferent renal component of the SNS can modulate central sympathetic outflow to the kidney, heart and vasculature in animals. The specific contribution of afferent nerve signalling in hypertension and in the potential antihypertensive effect of renal denervation has not been studied in humans.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* capable of discernment

Exclusion Criteria:

* having contra-indications for MRI (claustrophobia, cardiac pacemaker or other metallic or mechanical implant or device, etc.)
* pregnant women
* lower limb sensitive neuropathy
* Blood pressure >180/110 mmHg during washout period (for hypertensive patients)
* Intolerance to Sonovue®(ultrasound contrast agent)
* Acute or chronic disease other than hypertension that influences renal function
* taking medication/drugs, except of calcium channel blockers for resistant hypertensive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normotensive participants: university employees mainly Hypertensive patients: from the outpatient clinic of the Nephrology Service Resistant hypertensive patients (renal denervated and non-denervated): from the outpatient clinic of the Nephrology Service
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Change in brain BOLD signal intensity | 1.5 hours
  Changes in the brain BOLD fMRI signal of the brainstem in response to a cold pressor test

SECONDARY OUTCOMES:
Functional connectivity (resting state and effective connectivity) | 1.5 hours
  Activation patterns in spatially separated brain regions tending to have synchronous activity in resting state and activation pattern changes during a cold pressor test
Structural connectivity | 30 minutes
  Map of anatomical (neural) connections within the brain in normotensive subjects and hypertensive patients
Correlation between brain BOLD fMRI and renal ultrasound | 2 hours
  Correlation between changes in brain BOLD signal and renal (contrast-enhanced) ultrasound endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Wuerzner, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV, nephrology service, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data of participants that have signed the consent allowing their anonymized data to be shared, will be made available via the repository Zenodo
Supporting Information: Study Protocol, ICF
Time Frame: Once data are published
Access Criteria: available at zenodo :https://zenodo.org/
URL: https://zenodo.org/